CLINICAL TRIAL: NCT04487340
Title: Computer-based Online Database of Acute Stroke Patients for Stroke Management Quality Evaluation
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Shaoxing People's Hospital (Other); Affiliated Hospital of Jiaxing University (Other); Huzhou Center Hospital (Other); The Second Affiliated Hospital of Jiaxing University (Other); Jinhua Center Hospital (Unknown); Taizhou Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CASE II
Record Dates: First submitted 2020-07-19; First posted 2020-07-27 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Stroke, Acute
Keywords: thrombolysis; thrombectomy; hospitalization
MeSH Terms: conditions — Stroke | interventions — Educational Status

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Education — Provide each center with relevant education of guidelines, and help the clinicians to improve medical quality.

SUMMARY:
In the past three decades, the burden of stroke has increased in China and has gradually become the leading cause of death. The data acquisition and medical quality management still need to be improved in China. The purpose of this study was to establish online database of acute stroke patients for stroke management quality evaluation in China.

DETAILED DESCRIPTION:
This study is a prospective multi-center registration study. The data of acute ischemic stroke patients who underwent reperfusion therapy were registered on emergency platform. The data of stroke patients who were hospitalized were registered on stroke meidical quality control platform. The information including demographics, risk factors (history of hypertension, diabetes, stroke/TIA or atrial fibrillation, etc), prior antiplatelet usage, onset to door time (ODT), baseline National Institutes of Health Stroke Scale (NIHSS) score, baseline infarct core volume, laboratory data, ect were recorded. Clinical outcome at 3 months and 1 year was assessed.

ELIGIBILITY:
Inclusion Criteria:

Acute stroke patients

Exclusion Criteria:

No

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All acute stroke patients who were admitted to hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Independence (mRS 0-2) at 1 year | 1 year

SECONDARY OUTCOMES:
All-cause mortality at 1 year | 1 year
Brain hemorrhage at 24-72 hours after hospitalization | 72 hours
The incidence of recurrent stroke or other vascular events at 1 year | 1 year
Independence (mRS 0-2) at 5 year | 5 year
The incidence of recurrent stroke or other vascular events at 5 year | 5 year
All-cause mortality at 5 year | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Min Lou, PhD, Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Min Lou, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhou H, Zhong W, Zhang T, Xu C, Zhong G, Xie G, Zhang B, Chen H, Wang E, Xu D, Cheng C, Yang J, Lou M, Yan S; CASE-II Study Group. Comparing Outcomes of Thrombectomy Versus Intravenous Thrombolysis Based on Middle Cerebral Artery M2 Occlusion Features. Stroke. 2024 Jun;55(6):1592-1600. doi: 10.1161/STROKEAHA.123.044986. Epub 2024 May 24. PMID 38787930
- [Derived] Xue R, Zhong W, Zhou Y, He Y, Yan S, Chen Z, Wang J, Gong X, Lou M. Endovascular Treatment for Minor Acute Ischemic Strokes With Large Vessel Occlusion. J Am Heart Assoc. 2022 Dec 20;11(24):e027326. doi: 10.1161/JAHA.122.027326. Epub 2022 Dec 19. PMID 36533622
- [Derived] Wang J, Zhang J, Gong X, Zhang W, Zhou Y, Lou M. Prediction of large vessel occlusion for ischaemic stroke by using the machine learning model random forests. Stroke Vasc Neurol. 2022 Apr;7(2):94-100. doi: 10.1136/svn-2021-001096. Epub 2021 Oct 26. PMID 34702747